CLINICAL TRIAL: NCT00003468
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Children With Low Grade Astrocytoma
Brief Title: Antineoplaston Therapy in Treating Children With Low-Grade Astrocytoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066504; BC-BT-13 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2017-07

CONDITIONS: Low Grade Astrocytomas
Keywords: childhood low-grade astrocytoma; recurrent childhood astrocytoma; persistent childhood astrocytoma
MeSH Terms: interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a low grade astrocytoma that have not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for children with low grade astrocytomas that have not responded to standard therapy provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of children with low grade astrocytomas that have not responded to standard therapy

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children (> 6 months of age) with low grade astrocytomas that has not responded to standard therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with low grade gliomas that has not responded to standard therapy, as measured by an objective response to therapy (complete response, partial response or stable disease).
* To determine the safety and tolerance of Antineoplaston therapy in children with a brain tumor.

OVERVIEW: This is a single arm, open-label study in which children with low grade astrocytomas that have not responded to standard therapy receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed low grade astrocytoma.
* Evidence of persistent or progressive tumor after standard therapy by MRI scan performed within 2 weeks prior to study entry
* Tumor must be at least 5 mm

PATIENT CHARACTERISTICS:

Age:

* 6 months to 17 years

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 2,000/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension
* No history of congestive heart failure
* No other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids for cerebral edema allowed (must be on stable dose for at least 1 week prior to study entry)

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No prior antineoplaston therapy

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 1996-07; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski, SR, Janicki, TJ, Burzynski, G.S. A Phase II Study of Antineoplastons A10 and AS2-1 in Children with Low-Grade Astrocytomas-Final Report (Protocol BT-13). Submitted to Journal of Cancer Therapy, 2016
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eleven patients were recruited between July 1996 and November 2005. All study subjects were seen at the Burzynski Clinic in Houston TX
Groups:
- Antineoplaston Therapy: Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Children with a low-grade astrocytoma who have not responded to standard therapy will receive Antineoplaston therapy (Atengenal + Astugenal).
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 11
Completed | 9 (Two patients were not evaluable.)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: Years] | 9.3 [3.7 to 17.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks..
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 9
Participants
  Complete Response | 4
  Partial Response | 1
  Stable Disease | 4
  Progressive Disease | 0

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months overall survival
Time Frame: 6 months, 12 months, 24 months, 36 months, 48 months, 60 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 11
Percentage of participants
  6 months overall survival | 81.8
  12 months overall survival | 81.8
  24 months overall survival | 63.6
  36 months overall survival | 63.6
  48 months overall survival | 63.6
  60 months overall survival | 63.6

ADVERSE EVENTS:
Time Frame: 9 years, 6 months
Description: Adverse event data was collected through regular patient assessment and regular laboratory testing
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 6/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=11)
Central venous catheter infection (Infections and infestations) | 1 — The Central venous catheter infection was not related to Antineoplaston therapy.
Fever (General disorders) | 1 — The Fever was not related to Antineoplaston therapy.
Chicken pox (Infections and infestations) | 1 — The chicken pox was not related to Antineoplaston therapy.
Hypernatremia (Investigations) | 1 — The Hypernatremia was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 4 — The Seizures were not related to Antineoplaston therapy.
Pain: Abdomen NOS (Gastrointestinal disorders) | 1 — The Pain: Abdomen NOS was not related to Antineoplaston therapy.
Renal/Genitourinary-Other: kidney stones (Renal and urinary disorders) | 1 — The Renal/Genitourinary-Other: kidney stones were not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=11)
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 4
Allergic rhinitis (including sneezing, nasal stuffiness, 2 2 (General disorders) | 2
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 8
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4
Platelets (Blood and lymphatic system disorders) | 1
Supraventricular and nodal arrhythmia: Sinus bradycardia (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia: Sinus tachycardia (Cardiac disorders) | 2
Central venous catheter infection (Infections and infestations) | 5
Non-functional central venous cateter (General disorders) | 4
Pain : Central venous catheter (General disorders) | 1
Central venous catheter: Thrombosis/embolism (General disorders) | 1
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1
Constitutional Symptoms - Other (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 8
Fever (General disorders) | 5
Obesity (General disorders) | 1
Rigors/chills (General disorders) | 3
Weight gain (General disorders) | 5
Weight loss (General disorders) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2
Striae (Skin and subcutaneous tissue disorders) | 1
Edema/Fluid retention (General disorders) | 8
Cushingoid (Endocrine disorders) | 1
Cushingoid appearance (Endocrine disorders) | 4
Endocrine - Other (Endocrine disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 3
Anorexia (Gastrointestinal disorders) | 2
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 8
Distension/bloating, abdominal (Gastrointestinal disorders) | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 6
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Hemorrhage, GU: Urinary NOS (Renal and urinary disorders) | 3
Chicken pox (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 4
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1
Infection (documented clinically): Middle ear (otitis) (Infections and infestations) | 2
Infection (documented clinically): Blood (Infections and infestations) | 1
Infection (documented clinically): Pharynx (Infections and infestations) | 2
Infection (documented clinically): Sinus (Infections and infestations) | 2
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1
Albumin, serum-low (hypoalbuminemia) (Investigations) | 2
Alkaline phosphatase (Investigations) | 2
Bicarbonate, serum-low (Investigations) | 3
Hypercholesterolemia (Investigations) | 6
Hyperglycemia (Investigations) | 8
Hyperkalemia (Investigations) | 2
Hypernatremia (Investigations) | 9
Hypertriglyceridemia (Investigations) | 2
Hyperuricemia (Investigations) | 1
Hypocalcemia (Investigations) | 3
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 9
Hypomagnesemia (Investigations) | 3
Hyponatremia (Investigations) | 3
Hypophosphatemia (Investigations) | 3
Metabolic/Laboratory - Other (Investigations) | 5
Proteinuria (Investigations) | 4
SGOT (Investigations) | 5
SGPT (Investigations) | 6
Uric acid, serum-high (hyperuricemia) (Investigations) | 3
Muscle weakness: Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness: Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 3
Confusion (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 7
Memory impairment (Nervous system disorders) | 1
Mood alteration: Agitation (Nervous system disorders) | 1
Mood alteration: Depression (Nervous system disorders) | 1
Neurology - Other (Nervous system disorders) | 2
Neuropathy - cranial (Nervous system disorders) | 1
Neuropathy: CN III Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 4
Somnolence/depressed level of consciousness (Nervous system disorders) | 7
Speech impairment (Nervous system disorders) | 2
Syncope (fainting) (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 3
Vision-blurred vision (Eye disorders) | 2
Vision-flashing lights/floaters (Eye disorders) | 1
Vision-photophobia (Eye disorders) | 1
Pain: Abdomen NOS (Gastrointestinal disorders) | 3
Pain: Back (Musculoskeletal and connective tissue disorders) | 4
Pain: Buttock (Musculoskeletal and connective tissue disorders) | 1
Pain: Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 2
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain: Head/headache (Nervous system disorders) | 7
Pain: Joint (Musculoskeletal and connective tissue disorders) | 5
Pain: Lymph node (Blood and lymphatic system disorders) | 1
Pain: Muscle (Musculoskeletal and connective tissue disorders) | 2
Pain: Neck (Musculoskeletal and connective tissue disorders) | 3
Pain: Scalp (Skin and subcutaneous tissue disorders) | 1
Pain: Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pain: Urethra (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Renal/Genitourinary-Other: kidney stones (Renal and urinary disorders) | 1
Renal/Genitourinary-Other (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 7
Vascular - Other (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No